CLINICAL TRIAL: NCT03940196
Title: ENGOT-ov50 / GOG-3029 / INNOVATE-3: Pivotal, Randomized, Open-label Study of Tumor Treating Fields (TTFields, 200kHz) Concomitant With Weekly Paclitaxel for the Treatment of Recurrent Ovarian Cancer
Brief Title: Effect of Tumor Treating Fields (TTFields, 200 kHz) Concomitant With Weekly Paclitaxel for the Treatment of Recurrent Ovarian Cancer (ENGOT-ov50 / GOG-3029 / INNOVATE-3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF-28
Record Dates: First submitted 2019-04-29; First posted 2019-05-07 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Ovarian Cancer
Keywords: Platinum Resistant Ovarian Cancer; TTFields; Paclitaxel; Minimal toxicity; TTF; Tumor Treating Fields; Novocure
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- NovoTTF-100L(O) (Experimental): Patients receive TTFields using the NovoTTF-100L(O) System together with weekly Paclitaxel
  Interventions: Device: NovoTTF-100L(O); Drug: Paclitaxel
- Best Standard of Care (Active Comparator): Patients receive best standard of care with weekly Paclitaxel
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Device: NovoTTF-100L(O) — Patients receive continuous TTFields treatment using the NovoTTF-100L(O) device. TTFields treatment will consist of wearing four electrically insulated electrode arrays on the abdomen/pelvis. The treatment enables the patient to maintain regular daily routine.
  Other Names: TTFields
  Arms: NovoTTF-100L(O)
Drug: Paclitaxel — Paclitaxel 80 mg/m^2 intravenous infusion will be administered weekly for 8 weeks and then on Days 1, 8 and 15 of each subsequent 28-day cycle.
  Other Names: Weekly Paclitaxel; Taxol

SUMMARY:
The study is a prospective, randomized controlled phase III trial aimed to test the efficacy and safety of Tumor Treating Fields (TTFields) concomitant with weekly paclitaxel for the treatment of recurrent ovarian cancer . The device is an experimental, portable, battery operated device for chronic administration of alternating electric fields (termed TTFields or TTF) to the region of the malignant tumor, by means of surface, insulated electrode arrays.

DETAILED DESCRIPTION:
PAST PRE-CLINICAL AND CLINICAL EXPERIENCE:

The effect of the electric fields (TTFields, TTF) has demonstrated significant activity in in vitro and in vivo ovarian carcinoma pre-clinical models both as a single modality treatment and in combination with chemotherapies. TTFields have been demonstrated to act synergistically with taxanes and have been shown to be additive when combined with other chemotherapies. In addition, TTFields have shown to inhibit metastatic spread of malignant melanoma in in vivo experiment.

In a pilot study, 31 patients with recurrent platinum-resistant ovarian carcinoma received paclitaxel together with TTFields (200 kHz) applied to the abdomen/pelvis until disease progression. The combination was well tolerated and the only device-related adverse event was contact dermatitis.

In addition, a phase III trial of Optune® (200 kHz) as monotherapy compared to active chemotherapy in recurrent glioblastoma patients showed TTFields to be equivalent to active chemotherapy in extending survival, associated with minimal toxicity, good quality of life, and activity within the brain (14% response rate). Finally, a phase III trial of Optune® combined with maintenance temozolomide compared to maintenance temozolomide alone has shown that combined therapy led to a significant improvement in both progression free survival and overall survival in patients with newly diagnosed glioblastoma without the addition of high grade toxicity and without decline in quality of life.

DESCRIPTION OF THE TRIAL:

All patients included in this trial are patients with platinum-resistant ovarian carcinoma. In addition, all patients must meet all eligibility criteria.

Eligible patients will be randomly assigned to one of two groups:

1. Patients receive TTFields at 200 kHz to the abdomen and pelvis using the NovoTTF-100L(O) System together with weekly paclitaxel.
2. Patients receive weekly paclitaxel alone.

Patients will be randomized at a 1:1 ratio. Baseline tests will be performed in patients enrolled in both arms. If assigned to the NovoTTF-100L(O) group, the patients will be treated continuously with the device until progression in the abdomen/pelvis. On both arms, patients who have progression outside the abdomen/pelvis will switch to a second line treatment according to local practice.

SCIENTIFIC BACKGROUND:

Electric fields exert forces on electric charges similar to the way a magnet exerts forces on metallic particles within a magnetic field. These forces cause movement and rotation of electrically charged biological building blocks, much like the alignment of metallic particles seen along the lines of force radiating outwards from a magnet.

Electric fields can also cause muscles to twitch and if strong enough may heat tissues. TTFields are alternating electric fields of low intensity. This means that they change their direction repetitively many times a second. Since they change direction very rapidly (200 thousand times a second), they do not cause muscles to twitch, nor do they have any effects on other electrically activated tissues in the body (brain, nerves and heart). Since the intensities of TTFields in the body are very low, they do not cause heating.

The finding made by Novocure was that finely tuned alternating fields of very low intensity, now termed TTFields (Tumor Treating Fields), cause a significant slowing in the growth of cancer cells. Due to the unique geometric shape of cancer cells when they are multiplying, TTFields cause electrically-charged cellular components of these cells to change their location within the dividing cell, disrupting their normal function and ultimately leading to cell death. In addition, cancer cells also contain miniature building blocks which act as tiny motors in moving essential parts of the cells from place to place. TTFields interfere with the normal orientation of these tiny motors related to other cellular components since they are electrically-charged as well. As a result of these two effects, tumor cell division is slowed, results in cellular death or reverses after continuous exposure to TTFields.

Other cells in the body (normal healthy tissues) are affected much less than cancer cells since they multiply at a much slower rate if at all. In addition TTFields can be directed to a certain part of the body, leaving sensitive areas out of their reach. Finally, the frequency of TTFields applied to each type of cancer is specific and may not damage normally dividing cells in healthy tissues.

In conclusion, TTFields could potentially become treatment for ovarian cancer with very few side effects.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older
2. Epithelial histology of ovarian/primary peritoneal or fallopian tube carcinoma at the time of diagnosis
3. Life expectancy of ≥ 12 weeks
4. Maximum two prior lines of systemic therapy following diagnosis of platinum-resistance
5. Maximum total of 5 prior lines of systemic therapy
6. Amenable to receive weekly paclitaxel and able to operate the NovoTTF-100L(O) System
7. ECOG 0-1
8. Evaluable (measurable or non-measurable) disease in the abdominal/pelvic region per RECIST V1.
9. Signed informed consent form for the study protocol

Exclusion Criteria:

1. Primary platinum-refractory disease (progression per RECIST V1.1 during or within 1 month after first line therapy), while secondary platinum-refractory disease is allowed
2. Prior disease progression on a weekly paclitaxel for recurrent disease
3. Brain metastasis or leptomeningeal spread of the tumor
4. Albumin level <25 gram/liter (subjects should not receive total parenteral nutrition or albumin within 2 weeks of the test)
5. CTCAE V5.0 Grade 3 or higher peripheral neuropathy
6. Implantable electrical medical devices
7. Known allergies to medical adhesives or hydrogel
8. Known immediate or delayed hypersensitivity reaction or idiosyncrasy to paclitaxel or drugs similar or related to paclitaxel, except for cases that were able to undergo desensitization per investigator
9. Prior malignancies treated primarily or for recurrence within 2 years prior to inclusion in this study, except for completely resected non-melanomatous skin carcinoma, or successfully treated in situ carcinoma of the skin, breast or cervix of the uterus
10. Serious co-morbidities
11. Concurrent anti-tumor therapy beyond weekly paclitaxel, excluding hormonal therapy for breast cancer
12. Concurrent active treatment in another clinical trial. However prior participation in clinical trials is allowed as well as participation during survival follow-up
13. Pregnancy or breast-feeding (female patients with reproductive potential and their partners must accept to use effective contraception throughout the entire study period and for 3 months after the end of treatment). All patients who are capable of becoming pregnant must take a pregnancy test which is negative within 72 hours before beginning treatment. The definition of effective contraception is left up to the decision of the investigator
14. Admitted to an institution by administrative or court order

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Overall survival | 4 years

SECONDARY OUTCOMES:
Progression-free survival | 4 years
Objective response rate | 4 years
Next progression-free survival | 4 years
  Measured from the time of randomization to tumor progression on next-line treatment
Time to undisputable deterioration in health-related quality of life (HRQoL) | 4 years
  Measured as the time interval between randomization until the first decrease in HRQoL score ≥ 10-point with no further improvement in HRQoL score ≥ 10 points on any further HRQoL data, based on the EORTC QLQ-C30 questionnaire
Time to first and second subsequent treatment | 4 years
  Measured as the time from the date of randomization to the clinical decision made by the investigator to initiate a first and second subsequent lines of treatment, respectively, or death date
Quality of life using the EORTC QLQ C30 questionnaire with the ovarian cancer symptom OV28 module. | 4 years
Severity and frequency of adverse events | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ignace Vergote, MD, Principal Investigator — University Hospitals Leuven, Leuven Cancer Institute
Locations (118):
- United States (58):
  - Arizona Oncology- Biltmore Cancer Center, Phoenix, Arizona
  - Arizona Oncology, Tucson, Arizona
  - University of California, La Jolla, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - California Pacific Medical Center- Pacific Campus, San Francisco, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - University of Colorado Denver, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers, Longmont, Colorado
  - Rocky Mountain Cancer Centers, Parker, Colorado
  - Rocky Mountain Cancer Centers, Pueblo, Colorado
  - Rocky Mountain Cancer Centers, Thornton, Colorado
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - AdventHealth Cancer Institute, Orlando, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Rush University Cancer Center - Chicago and Innovation, Chicago, Illinois
  - Des Moines Oncology Research Association, Des Moines, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - Maryland Oncology Hematology, P.A., Silver Spring, Maryland
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Minnesota Oncology Hematology, PA, Saint Paul, Minnesota
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center of Hope at Renown Medical Center, Reno, Nevada
  - MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - The Valley Hospital, Paramus, New Jersey
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Miami Valley Hospital South, Centerville, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Northwest Cancer Specialists, PC, Portland, Oregon
  - West Penn OB/GYN, Pittsburgh, Pennsylvania
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Abington Hospital- Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Sanford Gynecologic Oncology Clinic, Sioux Falls, South Dakota
  - Texas Oncology Austin-Balcones, Austin, Texas
  - Texas Oncology Austin-Midtown, Austin, Texas
  - Texas Oncology Austin-North Austin, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Oncology, Dallas, Texas
  - Texas Oncology-Fort Worth, Fort Worth, Texas
  - The University of Texas Medical School at Houston, Houston, Texas
  - Texas Oncology-McAllen, McAllen, Texas
  - Texas Oncology San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology - Sugar Land, Sugar Land, Texas
  - Texas Oncology, The Woodlands, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Texas Oncology-Deke Slayton Cancer Center, Webster, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Carilion Clinic-Gynecologic Oncology, Roanoke, Virginia
  - Multicare Institute for Research and Innovation, Tacoma, Washington
- Austria (4):
  - KH der Barmherzigen Brüder Graz, Graz
  - Univ.-Klinik für Gynäkologie und Geburtshilfe, Graz
  - Univ.-Klinik für Gynäkologie und Geburtshilfe, Innsbruck, Innsbruck
  - Landesfrauenklinik Salzburg, Salzburg
- Belgium (8):
  - Imelda Ziekenhuis Bonheiden, Bonheiden
  - Cliniques Universitaires Saint Luc, Institut Roi Albert II, Brussels
  - Grand Hôpital de Charleroi, Oncologie-Hématologie, Charleroi
  - AZ Maria Middelares, Clinical Trial Unit Medical Oncology - Integrated Cancer Center Ghent, Ghent
  - UZ Gent, Ghent
  - University Hospitals Leuven, Leuven Cancer Institute, Leuven
  - CHU Ambroise Paré, Mons
  - CHU UCL Namur - Site Ste Elisabeth, Namur
- Canada (5):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Centre Hospitalie, Montreal, Quebec
  - Tom Baker Cancer Center, Calgary
  - McGill University Health Centre, Montreal
  - Jewish General Hospital, Montreal
- Czechia (5):
  - Gynekologicko-porodnické oddělení - Nemocnice České Budějovice a.s., České Budějovice
  - Onkologická Klinika Fakultní nemocnice Olomouc, Olomouc
  - University Hospital Ostrava, Ostrava-Poruba
  - Gynekologicko-porodnická klinika, Fakultní nemocnice Královské Vinohrady, Prague
  - Gynekologicko-porodnická klinika 1. LF UK a VFN, Prague
- Germany (3):
  - Charité Universitätsmedizin Berlin, Campus Virchow-Klinikum, Klinik für Gynäkologie, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Horst-Schmidt-Kliniken, Gynecology and Gynecologic, Oncology Department, Wiesbaden
- Hungary (3):
  - Semmelweis University, Budapest
  - Nőgyógyászati Osztály, Országos Onkológiai Intézet, Budapest
  - Szuleszeti és Nogyogyaszati Klinika, Debrecen
- Israel (4):
  - Hillel Yaffe Medical Center, Hadera
  - Saare Zedek Medical Center - Gyneco-Oncology, Jerusalem
  - Oncology Institute, Galilee Medical Center, Nahariya
  - Gyneco-Oncology Chaim Sheba Medical Center, Ramat Gan
- Italy (8):
  - Policlinico S. Orsola-Malpighi, SSD Oncologia Medica Addarii, Bologna
  - Presidio Ospedaliero Antonio Perrino - ASL Brindisi, Brindisi
  - ASST Lecco - Ospedale Manzoni, Dipartimento Oncologico, Lecco
  - Dipartimento Medicina e Chirurgia, Università Milano-Bicocca, Direttore Programma Ginecologia Oncologica, Istituto Europeo Oncologia, Milan
  - IRCCS Ospedale San Raffaele, U.O. Ginecologia-Ematologia e TMO, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Fondazione Policlinico Universitario Gemelli, Roma
  - University Saint Anna, Torino
- Netherlands (2):
  - Amsterdam Universitair Medische centra, Amsterdam
  - University Medical Center Utrech, Utrecht
- Poland (7):
  - Szpitale Pomorskie Sp. z o.o., Gdynia
  - Oddział Kliniczny Chirurgii Ogólnej i Onkologicznej, Szpital Św. Rafała, Krakow
  - Uniwersytet Medyczny w Lublinie, I Klinika Ginekologii Onkologicznej i Ginekologii, Lublin
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej MSWiA z Warmińsko-Mazurskim Centrum Onkologii w Olsztynie, Oddział Kliniczny Onkologii i Immunoonkologii z Ośrodkiem Dziennym Terapii Onkologicznej, Olsztyn
  - Oddział Ginekologii Onkologicznej Katedry i Kliniki Onkologii Uniwersytetu Medycznego w Poznaniu, Poznan
  - Samodzielny Publiczny Szpital Kliniczny Nr 2 PUM w Szczecinie, Klinika Ginekologii Operacyjnej i Onkologii Ginekologicznej Dorosłych i Dziewcząt, Szczecin
  - Szpital Kliniczny im. ks. Anny Mazowieckiej, Warsaw
- Spain (7):
  - Servicio de Oncología Médica, Hospital Universitario Quirón Dexeus, Barcelona
  - lnstitut Catala d'Oncologia, Hospital Universitario Dr. Josep Trueta, Servicio de Oncologia,, Girona
  - Clinica Universidad de Navarra en Madrid, Madrid
  - Hospital MD Anderson Cancer Center, Madrid
  - Hospital Universitario Ramon y Cajal, Servicio de Oncologia Médica, Madrid
  - Hospital 12 de Octubre. Servicio Oncología Médica, Madrid
  - Fundació Institut d'Investigació Sanitària Illes Balears - IdISBa, Hospital Universitari Son Espases, Palma de Mallorca
- Switzerland (4):
  - Gynecological Tumor Center, University Hospital Basel, Basel
  - IOSI Bellinzona, Oncology Institute of Southern Switzerland, Ospedale San Giovanni, Bellinzona
  - Kantonsspital Frauenfeld - Frauenklinik, Frauenfeld
  - UniversitätsSpital Zürich - Klinik für Gynäkologie, Zurich

REFERENCES:
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Stupp R, Wong ET, Kanner AA, Steinberg D, Engelhard H, Heidecke V, Kirson ED, Taillibert S, Liebermann F, Dbaly V, Ram Z, Villano JL, Rainov N, Weinberg U, Schiff D, Kunschner L, Raizer J, Honnorat J, Sloan A, Malkin M, Landolfi JC, Payer F, Mehdorn M, Weil RJ, Pannullo SC, Westphal M, Smrcka M, Chin L, Kostron H, Hofer S, Bruce J, Cosgrove R, Paleologous N, Palti Y, Gutin PH. NovoTTF-100A versus physician's choice chemotherapy in recurrent glioblastoma: a randomised phase III trial of a novel treatment modality. Eur J Cancer. 2012 Sep;48(14):2192-202. doi: 10.1016/j.ejca.2012.04.011. Epub 2012 May 18. PMID 22608262
- [Background] Kirson ED, Giladi M, Gurvich Z, Itzhaki A, Mordechovich D, Schneiderman RS, Wasserman Y, Ryffel B, Goldsher D, Palti Y. Alternating electric fields (TTFields) inhibit metastatic spread of solid tumors to the lungs. Clin Exp Metastasis. 2009;26(7):633-40. doi: 10.1007/s10585-009-9262-y. Epub 2009 Apr 23. PMID 19387848
- [Background] Giladi M, Schneiderman RS, Voloshin T, Porat Y, Munster M, Blat R, Sherbo S, Bomzon Z, Urman N, Itzhaki A, Cahal S, Shteingauz A, Chaudhry A, Kirson ED, Weinberg U, Palti Y. Mitotic Spindle Disruption by Alternating Electric Fields Leads to Improper Chromosome Segregation and Mitotic Catastrophe in Cancer Cells. Sci Rep. 2015 Dec 11;5:18046. doi: 10.1038/srep18046. PMID 26658786
- [Background] Stupp R, Taillibert S, Kanner AA, Kesari S, Steinberg DM, Toms SA, Taylor LP, Lieberman F, Silvani A, Fink KL, Barnett GH, Zhu JJ, Henson JW, Engelhard HH, Chen TC, Tran DD, Sroubek J, Tran ND, Hottinger AF, Landolfi J, Desai R, Caroli M, Kew Y, Honnorat J, Idbaih A, Kirson ED, Weinberg U, Palti Y, Hegi ME, Ram Z. Maintenance Therapy With Tumor-Treating Fields Plus Temozolomide vs Temozolomide Alone for Glioblastoma: A Randomized Clinical Trial. JAMA. 2015 Dec 15;314(23):2535-43. doi: 10.1001/jama.2015.16669. PMID 26670971
- [Background] Stupp R, Taillibert S, Kanner A, Read W, Steinberg D, Lhermitte B, Toms S, Idbaih A, Ahluwalia MS, Fink K, Di Meco F, Lieberman F, Zhu JJ, Stragliotto G, Tran D, Brem S, Hottinger A, Kirson ED, Lavy-Shahaf G, Weinberg U, Kim CY, Paek SH, Nicholas G, Bruna J, Hirte H, Weller M, Palti Y, Hegi ME, Ram Z. Effect of Tumor-Treating Fields Plus Maintenance Temozolomide vs Maintenance Temozolomide Alone on Survival in Patients With Glioblastoma: A Randomized Clinical Trial. JAMA. 2017 Dec 19;318(23):2306-2316. doi: 10.1001/jama.2017.18718. PMID 29260225
- [Background] Vergote I, von Moos R, Manso L, Van Nieuwenhuysen E, Concin N, Sessa C. Tumor Treating Fields in combination with paclitaxel in recurrent ovarian carcinoma: Results of the INNOVATE pilot study. Gynecol Oncol. 2018 Sep;150(3):471-477. doi: 10.1016/j.ygyno.2018.07.018. Epub 2018 Jul 27. PMID 30060963
- [Background] Taphoorn MJB, Dirven L, Kanner AA, Lavy-Shahaf G, Weinberg U, Taillibert S, Toms SA, Honnorat J, Chen TC, Sroubek J, David C, Idbaih A, Easaw JC, Kim CY, Bruna J, Hottinger AF, Kew Y, Roth P, Desai R, Villano JL, Kirson ED, Ram Z, Stupp R. Influence of Treatment With Tumor-Treating Fields on Health-Related Quality of Life of Patients With Newly Diagnosed Glioblastoma: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2018 Apr 1;4(4):495-504. doi: 10.1001/jamaoncol.2017.5082. PMID 29392280